CLINICAL TRIAL: NCT03336528
Title: A Randomized Controlled Trial Comparing Insulin Degludec and Glargine U100 for the Inpatient and Post-Hospital Discharge Management of Medicine and Surgery Patients With Type 2 Diabetes
Brief Title: Insulin Degludec and Glargine U100 for Management of Hospitalized and Discharged Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Guillermo Umpierrez, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00087816
Record Dates: First submitted 2017-11-06; First posted 2017-11-08 (Actual); Results first posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Type 2 Diabetes
Keywords: Long-acting insulin analog
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin degludec; Insulin Glargine; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Degludec inpatient (Experimental): Study participants treated with insulin prior to admission will receive 80% or 100% of the total daily dose (TDD) given as a basal bolus regimen with degludec once daily plus rapid-acting aspart insulin before meals.
  Interventions: Drug: Degludec; Drug: Aspart
- Glargine U100 inpatient (Active Comparator): Study participants treated with insulin prior to admission will receive 80% or 100% of the total daily dose (TDD) given as basal bolus regimen with glargine once daily plus rapid-acting aspart insulin before meals.
  Interventions: Drug: Glargine; Drug: Aspart

INTERVENTIONS:
Drug: Degludec — Degludec is a long-acting human insulin analog indicated to improve glycemic control in adults with diabetes mellitus. Patients will be treated with bolus regimen given half of total daily dose (TDD) as basal once daily and half as aspart divided in three equal doses before meals. Patients with poor oral intake or with medical instruction to withhold oral intake (NPO) will receive the basal dose, but prandial dose will be held. Insulin dose will be adjusted daily to maintain a fasting and pre-dinner blood glucose (BG) between 100 mg/dL and 180 mg/dL.
  Other Names: Tresiba
  Arms: Degludec inpatient
Drug: Glargine — Glargine is a long-acting human insulin analog indicated to improve glycemic control in adults with diabetes mellitus. Patients will be treated with bolus regimen given half of total daily dose (TDD) as basal once daily and half as aspart divided in three equal doses before meals. Patients with poor oral intake or with medical instruction to withhold oral intake (NPO) will receive the basal dose, but prandial dose will be held. Insulin dose will be adjusted daily to maintain a fasting and pre-dinner BG between 100 mg/dL and 180 mg/dL.
  Other Names: Lantus
  Arms: Glargine U100 inpatient
Drug: Aspart — Aspart insulin will be given in three equally divided doses before each meal. To prevent hypoglycemia, if a subject is not able to eat, aspart insulin dose will be held.
  Other Names: Novolog

SUMMARY:
The purpose of this study is to find out if treatment with degludec insulin when compared to glargine U100 insulin will result in similar blood sugar control in patients with diabetes who are admitted to the hospital and then transition to home after discharge from the hospital.

DETAILED DESCRIPTION:
Degludec is a new generation basal insulin analog with a longer duration of action compared to insulin glargine. Several outpatient trials have reported that treatment with degludec results in comparable improvement in HbA1c levels and in lower rates of hypoglycemia compared to glargine U100 insulin. However, no previous studies have compared the safety and efficacy of the long-acting basal insulin degludec in the inpatient management of patients with diabetes. It is expected that a large number of patients with diabetes will be started on or transitioned to this new insulin formulation so acquiring knowledge on the safety and efficacy of degludec insulin is of great clinical interest. Accordingly, the proposed study will provide novel and clinically useful information on the efficacy (assessed as blood glucose control) and safety (assessed as hypoglycemia) of degludec in the inpatient setting and after hospital discharge in general medicine and surgery patients with Type 2 Diabetes (T2D).

Participants will be randomized to receive either a basal bolus with degludec or glargine U100 once daily during hospitalization. All participants will receive aspart insulin before meals. Participants with poorly controlled diabetes during the inpatient portion of the study will be invited to participate in the outpatient portion of the study. Participants in the outpatient portion of the study will be discharged on their preadmission oral antidiabetic medications plus degludec or glargine once daily, based on the study medication they were randomized to take during the inpatient portion of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females > 18 years of age who are admitted to a general medicine or surgical service
2. A known history of T2D treated either with diet alone, oral monotherapy, any combination of oral antidiabetic agents, short-acting glucagon-like peptide-1 receptor agonists (GLP-1 RA) or insulin therapy except for degludec and glargine U300
3. Subjects with diet alone and HbA1c>7.0%
4. Medical and surgical patients expected to be admitted length of stay (LOS) longer than 2 days
5. Subjects must have a randomization BG > 140 mg and < 400 mg/dL without laboratory evidence of diabetic ketoacidosis (bicarbonate < 18 milliequivalent (mEq)/L, potential of hydrogen (pH) < 7.30, or positive serum or urinary ketones)
6. Signed, informed consent and HIPAA documentation prior to any study procedures

Exclusion Criteria:

1. Subjects with increased BG concentration, but without a known history of diabetes (stress hyperglycemia)
2. Subjects treated with diet alone (no antidiabetic agents) and admission HbA1c <7%
3. Admission or pre-randomization BG≥400 mg/dL
4. Subjects with a history of diabetic ketoacidosis and hyperosmolar hyperglycemic state, or ketonuria
5. Patients treated with degludec or glargine U300, or with long-acting weekly GLP-1 RA (weekly exenatide, dulaglutide or albiglutide)
6. Patients with acute critical or surgical illness admitted to the ICU except for observation (<24 hours and did not require vasopressors and/or mechanical ventilation)
7. Patients with history of clinically relevant hepatic disease (diagnosed liver cirrhosis and portal hypertension), ongoing corticosteroid therapy (equal to a prednisone dose ≥5 mg/day), or impaired renal function (eGFR< 30 ml/min), or congestive heart failure (NYHA- IV)
8. Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study
9. Female subjects who are pregnant or breast feeding at time of enrollment into the study
10. Known or suspected allergy to trial medication(s), excipients, or related products
11. Previous participation in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Umpierrez, MD, Principal Investigator — Emory University
Locations (4):
- United States (4):
  - Grady Hospital, Atlanta, Georgia
  - Emory University Hospital Clinical Research Network, Atlanta, Georgia
  - Mount Sinai, New York, New York
  - Providence Medical Research Centre, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Yes
The research team will share individual participant data that underlie the results reported in this study, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available for sharing starting 6 months after publication and up to 5 years after publication.
Access Criteria: Access will be given to researchers who provide a methodologically sound proposal to achieve the aims in their approved proposal. Proposals should be directed to geumpie@emory.edu. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Result] Galindo RJ, Pasquel FJ, Vellanki P, Alicic R, Lam DW, Fayfman M, Migdal AL, Davis GM, Cardona S, Urrutia MA, Perez-Guzman C, Zamudio-Coronado KW, Peng L, Tuttle KR, Umpierrez GE. Degludec hospital trial: A randomized controlled trial comparing insulin degludec U100 and glargine U100 for the inpatient management of patients with type 2 diabetes. Diabetes Obes Metab. 2022 Jan;24(1):42-49. doi: 10.1111/dom.14544. Epub 2021 Sep 24. PMID 34490700

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from four study sites in the United States: Emory University Hospital and Grady Memorial Hospital in Atlanta, Georgia, Icahn School of Medicine at Mount Sinai in New York, New York, and Providence Medical Research Center in Spokane, Washington. Enrollment began on January 2, 2018 and all follow up was complete by March 1, 2021.
Groups:
- Degludec: Study participants randomized during hospitalization to receive 80% or 100% of their total daily dose (TDD) of outpatient insulin given as a basal bolus regimen with degludec once daily plus rapid-acting aspart insulin before meals.
  Degludec is a long-acting human insulin analog indicated to improve glycemic control in adults with diabetes mellitus. Participants were treated with an insulin regimen of half of TDD given a as basal insulin once daily and half as aspart divided in three equal doses before meals. Insulin dosage was adjusted daily to maintain a fasting and pre-dinner blood glucose between 100 and 180 mg/dL.
- Glargine: Study participants randomized during hospitalization to receive 80% or 100% of their total daily dose (TDD) of outpatient insulin given as basal bolus regimen with glargine once daily plus rapid-acting aspart insulin before meals.
  Glargine is a long-acting human insulin analog indicated to improve glycemic control in adults with diabetes mellitus. Participants were treated with an insulin regimen of half of TDD given as basal once daily and half as aspart divided in three equal doses before meals. Insulin dosage was adjusted daily to maintain a fasting and pre-dinner blood glucose between 100 and 180 mg/dL.
Period: Overall Study
Arm/Group | Degludec | Glargine
Started | 92 | 88
Participated in Optional Outpatient Study | 72 | 59
Completed (Completed inpatient portion of the study) | 82 | 79
Not Completed | 10 | 9
Not completed — Protocol Violation | 1 | 1
Not completed — Discharged within 48 hours of study medication | 8 | 6
Not completed — Did not receive study medication | 1 | 2

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes participants who completed the inpatient portion of the study and had at least two doses of the study medication.
Groups:
- Degludec: Study participants randomized during hospitalization to receive 80% or 100% of their total daily dose (TDD) of outpatient insulin given as a basal bolus regimen with degludec once daily plus rapid-acting aspart insulin before meals.
- Glargine: Study participants randomized during hospitalization to receive 80% or 100% of their total daily dose (TDD) of outpatient insulin given as basal bolus regimen with glargine once daily plus rapid-acting aspart insulin before meals.
- Total: Total of all reporting groups
Arm/Group | Degludec | Glargine | Total
Number analyzed (Participants) | 82 | 79 | 161
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.6 (12) | 56.7 (10) | 56.2 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 25 | 60
  Male | 47 | 54 | 101
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 10 | 18
  Not Hispanic or Latino | 74 | 69 | 143
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 58 | 56 | 114
  White | 16 | 18 | 34
  More than one race | 7 | 5 | 12
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 82 | 79 | 161
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 36 (9) | 36 (12) | 36 (11)
Home diabetes treatment [Count of Participants; unit: Participants]
  No treatment | 7 | 10 | 17
  Oral diabetic agents | 18 | 15 | 33
  Insulin only | 30 | 32 | 62
  Insulin plus oral diabetic agent | 27 | 21 | 48
  Glucagon-like peptide-1 receptor agonists (GLP-1RA) | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Daily Blood Glucose Concentration in Hospitalized Patients
Description: Blood glucose was measured before each meal and at bedtime among hospitalized study participants. Mean daily blood glucose concentration was calculated to determine differences in inpatient glycemic control in general medicine and surgery patients with Type 2 Diabetes (T2D) treated with basal bolus regimen with insulin degludec or glargine once daily plus aspart insulin before meals. A random (non-fasting) blood glucose measurement of 140 mg/dL or less is considered normal, while a measurement of 200 mg/dL or more indicates diabetes.
Time Frame: Baseline, up to the first 10 days of therapy
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Degludec | Glargine
Number analyzed (Participants) | 82 | 79
mg/dL
  Baseline | 219.50 (50.21) | 218.19 (54.56)
  Day 1 up to Day 10 | 179.75 (38.45) | 180.67 (45.10)

2. Primary Outcome: Mean Daily Blood Glucose Concentration in Discharged Patients.
Description: Blood glucose was measured before each meal and at bedtime, after participants were discharged from the hospital. Mean daily blood glucose concentration was calculated to determine differences in outpatient glycemic control in patients with Type 2 Diabetes (T2D) treated with basal bolus regimen with insulin degludec or glargine once daily plus aspart insulin before meals. Information was collected via bi-weekly phone interviews and during the outpatient study visits at Weeks 4 and 12.
Time Frame: Day after hospital discharge to 4 weeks after discharge, 4 to 12 weeks after hospital discharge
Population: This analysis includes participants completing the outpatient study visits.
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Degludec During Hospitalization: Study participants randomized during hospitalization to receive 80% or 100% of their total daily dose (TDD) of outpatient insulin given as a basal bolus regimen with degludec once daily plus rapid-acting aspart insulin before meals.
- Glargine During Hospitalization: Study participants randomized during hospitalization to receive 80% or 100% of their total daily dose (TDD) of outpatient insulin given as basal bolus regimen with glargine once daily plus rapid-acting aspart insulin before meals.
Arm/Group | Degludec During Hospitalization | Glargine During Hospitalization
Number analyzed (Participants) | 72 | 59
mg/dL
  Day after discharge up to the 4 week post-discharge study visit | 157.0 (46.4) | 143.0 (42.5)
  4 week post-discharge up to the 12 week post-discharge study visit | 148.7 (43.6) | 133.8 (44.2)

3. Secondary Outcome: Number of Blood Glucose Point-of-care Test Results Between 70 and 180 mg/dL in Hospitalized Patients
Description: Blood glucose was measured with point-of-care testing before each meal and at bedtime, and the count of blood glucose test results between 70 mg/dL and 180 mg/dL was determined.
Time Frame: During the first 10 days of therapy
Measure: Count of Units; unit: Blood Glucose Point-of-Care Test
Units Other Than Participants: Blood Glucose Point-of-Care Test
Arm/Group | Degludec | Glargine
Number analyzed (Participants) | 82 | 79
Number analyzed (Blood Glucose Point-of-Care Test) | 1378 | 1434
Blood Glucose Point-of-Care Test | 758 | 789

4. Secondary Outcome: Number of Participants With an Episode of Hypoglycemia While Hospitalized
Description: Blood glucose (BG) was measured before each meal and at bedtime. The number of participants with at least one hypoglycemic episode, defined as BG of 54 to 70 mg/dL, is presented here.
Time Frame: During the first 10 days of therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Degludec | Glargine
Number analyzed (Participants) | 82 | 79
Participants | 14 | 15

5. Secondary Outcome: Number of Participants With an Episode of Clinically Significant Hypoglycemia While Hospitalized
Description: Blood glucose was measured before each meal and at bedtime. The number of participants with at least one episode of clinically significant hypoglycemia, defined as BG < 54 mg/dL, is presented here.
Time Frame: During the first 10 days of therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Degludec | Glargine
Number analyzed (Participants) | 82 | 79
Participants | 3 | 1

6. Secondary Outcome: Number of Participants With an Episode of Severe Hypoglycemia While Hospitalized
Description: Blood glucose as measured before each meal and at bedtime. The number of participants with at least one episode of severe hypoglycemia, defined as BG < 40 mg/dL, is presented here.
Time Frame: During the first 10 days of therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Degludec | Glargine
Number analyzed (Participants) | 82 | 79
Participants | 0 | 0

7. Secondary Outcome: Number of Participants With an Episode of Severe Hyperglycemia While Hospitalized
Description: Blood glucose was measured before each meal and at bedtime. The number of participants who experienced at least one episode of severe hyperglycemia, defined as BG > 240 mg/dL, is presented here.
Time Frame: During the first 10 days of therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Degludec | Glargine
Number analyzed (Participants) | 82 | 79
Participants | 52 | 47

8. Secondary Outcome: Daily Dose of Insulin in Hospitalized Patients
Description: Electronic medical records and nursing records documented the day day and time of insulin administration, including the basal study drug given once daily (degludec or glargine), prandial insulin given before meals (aspart), and supplemental insulin given to correct hyperglycemia. The mean daily doses of basal insulin, prandial insulin, and total daily dose of insulin given to hospitalized patients are presented here.
Time Frame: During the first 10 days of therapy
Measure: Mean (Standard Deviation); unit: International Units of insulin
Arm/Group | Degludec | Glargine
Number analyzed (Participants) | 82 | 79
International Units of insulin
  Basal Insulin | 30 (13) | 30 (18)
  Prandial Insulin | 11 (9) | 12 (11)
  Total Daily Dose of Insulin | 56 (24) | 60 (36)

9. Secondary Outcome: Hemoglobin A1c (HbA1c) in Discharged Patients
Description: The HbA1C test reflects the average of a person's blood glucose levels over the past 3 months by measuring the percentage of red blood cells (RBCs) with glycated hemoglobin (hemoglobin with glucose bonded to it). Participants with HbA1C ≥ 7.5% were followed for 12 weeks after hospital discharge. Samples for HbA1C were drawn at 4 and 12 weeks post-discharge. An HbA1c measurement below 5.7% is considered normal, while a measurement of 6.5% or greater indicates diabetes.
Time Frame: 4 and 12 weeks after hospital discharge
Population: This analysis includes participants completing the outpatient study visits.
Measure: Mean (Standard Deviation); unit: percent of RBCs with glycated hemoglobin
Arm/Group | Degludec | Glargine
Number analyzed (Participants) | 72 | 59
percent of RBCs with glycated hemoglobin
  4 weeks post-discharge | 8.3 (1.4) | 8.0 (1.4)
  12 weeks post-discharge | 8.2 (1.9) | 7.4 (1.6)

10. Secondary Outcome: Number of Hypoglycemia Episodes in Discharged Patients
Description: Blood glucose was measured before each meal and at bedtime. The number of hypoglycemia episodes, defined as BG < 70 mg/dL, was recorded via bi-weekly phone interviews and during 4 and 12 week outpatient study visits.
Time Frame: Up to 12 weeks after hospital discharge
Population: This analysis includes participants completing the outpatient study visits.
Measure: Number; unit: episodes of hypoglycemia
Arm/Group | Degludec | Glargine
Number analyzed (Participants) | 72 | 59
episodes of hypoglycemia | 16 | 19

11. Secondary Outcome: Number of Clinically Significant Hypoglycemia Episodes in Discharged Patients
Description: Blood glucose will be measured before each meal and at bedtime. The number of episodes of clinically significant hypoglycemia, defined as BG < 54 mg/dL, are presented here.
Time Frame: Up to 12 weeks after hospital discharge
Population: This analysis includes participants completing the outpatient study visits.
Measure: Number; unit: episodes of significant hypoglycemia
Arm/Group | Degludec | Glargine
Number analyzed (Participants) | 72 | 59
episodes of significant hypoglycemia | 1 | 1

12. Secondary Outcome: Number of Episodes of Severe Hyperglycemia in Discharged Patients
Description: Blood glucose was measured before each meal and at bedtime. The number of episodes of severe hyperglycemia, defined as BG > 240 mg/dL, are presented here.
Time Frame: Up to 12 weeks after hospital discharge
Population: This analysis includes participants completing the outpatient study visits.
Measure: Number; unit: episodes of severe hyperglycemia
Arm/Group | Degludec | Glargine
Number analyzed (Participants) | 72 | 59
episodes of severe hyperglycemia | 211 | 55

13. Other Pre Specified Outcome: Number of Participants Experiencing Cardiac Complications During Hospitalization
Description: Cardiac complications during hospitalization were examined as a composite of complications, defined as myocardial infarction, cardiac arrhythmia requiring medical treatment, or cardiac arrest. The number of participants experiencing cardiac complications while hospitalized patients is presented here.
Time Frame: During the first 10 days of therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Degludec | Glargine
Number analyzed (Participants) | 82 | 79
Participants | 0 | 0

14. Other Pre Specified Outcome: Number of Participants With Acute Kidney Injury During Hospitalization
Description: Acute kidney injury defined as an increase in serum creatinine ≥ 0.3 mg/dL from baseline or ≥1.5 times baseline creatinine, per Kidney Disease: Improving Global Outcomes (KDIGO) guidelines. The number of participants experiencing acute kidney injury during hospitalization is presented here.
Time Frame: During the first 10 days of therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Degludec | Glargine
Number analyzed (Participants) | 82 | 79
Participants | 5 | 10

15. Other Pre Specified Outcome: Length of Hospital Stay
Description: The length of hospital in days is presented here.
Time Frame: Duration of hospital stay (an average of 10 days)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Degludec | Glargine
Number analyzed (Participants) | 82 | 79
days | 6.7 [4.7 to 10.5] | 7.5 [4.7 to 11.6]

16. Other Pre Specified Outcome: Number of Participants Who Died During Hospitalization
Description: Hospital mortality is evaluated as the number of deaths among participants during hospitalization.
Time Frame: Duration of hospital stay (an average of 10 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Degludec | Glargine
Number analyzed (Participants) | 82 | 79
Participants | 0 | 1

17. Other Pre Specified Outcome: Number of Participants Experiencing Acute Kidney Injury in Discharged Patients
Description: Acute kidney injury defined as an increase in serum creatinine ≥ 0.3 mg/dL from baseline or ≥1.5 times baseline creatinine, per Kidney Disease: Improving Global Outcomes (KDIGO) guidelines. The number of participants experiencing acute kidney injury after hospital discharge is presented here.
Time Frame: Up to 12 weeks after hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Degludec | Glargine
Number analyzed (Participants) | 72 | 59
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected from the time of consent during hospitalization for up to 3 months after hospital discharge.
Description: During hospitalization, electronic medical records were reviewed daily from the time of consent up to discharge. Any complication not present at the time of consent and that arose 48 hours after randomization was considered an adverse event. After discharge, participants were asked about any hospital readmissions and emergency room visits. Electronic medical records were also reviewed to document any hospital readmissions and emergency room visits among all study participants.
Arm/Group | Degludec | Glargine
All-Cause Mortality (participants affected / at risk) | 1/82 | 1/79
Serious Adverse Events (participants affected / at risk) | 3/82 | 3/79
Other Adverse Events (participants affected / at risk) | 3/82 | 3/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Degludec (N=82) | Glargine (N=79)
Hospital readmission for chest pain (Cardiac disorders) | 0 (0) | 1 (1)
Hospital readmission for urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1)
Hospital readmission for head injury (Nervous system disorders) | 0 (0) | 1 (1) — Head injury during rehabilitation resulting in coma
Hospital readmisson for non-healing amputation stump (Infections and infestations) | 1 (1) | 0 (0)
Hospital readmission for heart failure (Cardiac disorders) | 1 (3) | 0 (0)
Severe hypoglycemia (Endocrine disorders) | 1 (1) | 0 (0) — Hypoglycemia ≤ 40 mg/dL
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Degludec (N=82) | Glargine (N=79)
Emergency room visit for blunt chest trauma (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Emergency room visit for bilateral knee pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Emergency room visit for wound infection (Infections and infestations) | 1 (1) | 0 (0)
Emergency room visit for right eye medial stye (Eye disorders) | 0 (0) | 1 (1)
Emergency room visit for congestive heart failure (Cardiac disorders) | 1 (1) | 0 (0)
Emergency room visit for orthostatic hypotension (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-17): https://cdn.clinicaltrials.gov/large-docs/28/NCT03336528/Prot_SAP_000.pdf